**Document Name: Informed Consent Form** 

Date: 3 January 2023



## **Aalana Palana**

#### Section 1: PIS

# **Information Sheet for Caregiver-Child Dyads**

Greetings! I'm [ASSESSOR NAME] from Sangath. We are a non-governmental organization that has been working in the field of child development for the last 25 years. This interview is a part of an intervention called Aalana Palana developed by Sangath and UNICEF for promoting early child development. We are working closely with your local Anganwadi and would like to speak to pregnant women and mothers with children less than 3 years old.

<u>Instruction for assessor: Before proceeding further please ask the following.</u>

| Sno. | Item | Response Options | Variable Name |
|---|---|---|---|
| 1 | Is there a pregnant woman in the | Yes1 | |
| | house | No0 | |
| 2 | Is there a child in the house who has | Yes1 | |
| | not yet celebrated their 3 <sup>rd</sup> birthday? | No0 | |
| | If both 1 & 2 are "NO", thank the respondent and tell them that you will visit them again in a few | | |
| | months. | | |
| | END FORM | | |
| 3 | How many families are there in your | | |
| | household who have either a | | |
| | pregnant woman or a child who has | | |
| | not yet celebrated their 3 <sup>rd</sup> birthday? | | |
| | Note: each family is defined by a | | |
| | married couple or single parent and | | |
| | their children. | | |
| | Instruction: Separate consent & assessment forms will need to be generated for each family | | |
| mentioned in Q3. | | | |
| 4 | Is the pregnant woman or the | Yes1 | |
| | primary care giver of the child | No0 | |
| | available for the interview? | | |
| | If 4 is "NO" please ask for a suitable to | ime to revisit when the pregnant woman or | the primary care |
| | giver of the child will be available for the interview. Thank the respondent and plan revisit | | |
| | appropriately. | | |
| | END FORM. | | |

<u>Instruction for assessor: Share the PIS and administer the consent form ONLY to primary respondents</u> i.e., pregnant women and primary caregivers of children less than 3 years of age.

(Instruction to assessor: repeat the first paragraph if the first contact within the household was not a <u>primary respondent</u>) Greetings! I'm [ASSESSOR NAME] from Sangath. We are a non-governmental organization that has been working in the field of child development for the last 25 years. This interview is a part of an intervention called Aalana Palana developed by Sangath and UNICEF for

promoting early child development. We are working closely with your local Anganwadi and would like to speak to pregnant women and mothers with children less than 3 years old.

I would be grateful if you could assist me by participating in this interview. As I explain more about this, please feel free to ask questions or let me know if you need a break. In this interview, I will be asking you a few questions about your child and the type of things he/she can currently do. This interview will take approximately half an hour of your time. I would also like to come back to visit you every 3-4 months to do similar interviews.

There are no physical risks involved for you and your family if you agree to participate, although we will require you to give us your time for the same.

Your participation is entirely voluntary; this means that it is your choice whether to participate or not. There is no monetary compensation for participating in this interview. Even if you decide to participate now, you can change your mind in the middle of the interview and stop participating at any time. This will not influence any of the health and welfare—related services that you may be receiving.

Confidentiality is important to us. Any information taken from you will not be shared with anyone who is not part of the project team. Any identifiable information like your name, address, etc. that is collected during this interview will be stored safely, and only the team will be able to see it. After looking at all the information gathered, we may use it in presentations, reports and research papers. However, we will not mention any personal details that could identify you as a participant.

Do you have any questions?

If you have any questions you may ask them now or later, even after the interview has started. I will share our contact details with you, please do not hesitate to contact us.

# Shilpa Kasu

Sangath

UNICEF Office for Andhra Pradesh, Telangana & Karnataka

317/A, MLA Colony, Road No. 12, Banjara Hills,

Hyderabad - 500 034

Contact number: 07416317799

#### Ms Urvita Bhatia

Member Secretary, Sangath IRB,

Phone: +91 788 787 2345 Email: irb@sangath.in

## Gitanjali Lall

Sangath, Plot No. E5, Lane 1, 3rd & 4th Floor

Western Marg, Saiyad-Ul-Ajaib, Saket,

New Delhi 110030

## **Section 2: Consent Form**

#### **Consent Form for Caregiver-Child Dyad**

Script 1: 'Now I would request for your verbal consent. I will read out a few statements and ask for your consent on each. Your consent, or absent of it, will in no way interfere with any of the health and welfare-related services that you may be receiving.'

Instruction to Assessor: Please tick ( $\checkmark$ ) in the box

## A. Consent for Participation in Survey

# Aalana Palana Evaluations\_3 Jan 2023\_English

| 1 | I confirm that I have understood the information sheet and have had the opportunity to ask questions. | |
|---|---|---|
| 2 | I understand that my participation is voluntary and I will not receive any financial compensation for this. | |
| 3 | I am free to withdraw at any time without giving a reason and without affecting the benefits obtained from health & welfare-related schemes. | |
| 4 | I agree to take part in this interview. | |
| 5 | I understand that my personal data will be kept confidential. They will be reviewed by senior project staff but will not be shared outside of the project team. | |
| 6 | I agree for images and data taken during the sessions to be used by SANGATH and its partners for purposes of training, reports, websites, social media, national/international publications, and presentations in global conferences. | |
| Consent Status | | Consent Given |
| 7 | I agree to be visited once every 3-4 months to participate in similar interviews. (Optional) | |
| Name of Child: | | |
| Name of Primary Caregiver: | | |
| Name of Assessor: | | |
| Date: D D / M M M / Y Y Y | | |

Signature of Assessor

Signature of Parent/Caregiver